CLINICAL TRIAL: NCT07006207
Title: Deciphering Brain Olfactory Pathways in Prader-Willi Syndrome
Brief Title: Brain Olfactory Pathways in Prader-Willi Syndrome
Acronym: PRADOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0653
Record Dates: First submitted 2025-05-13; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Prader-Willi Syndrome
Keywords: cerebral activity; Olfactory activation
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT exposed patients (Experimental): children OT exposed have olfactory test and fMRI
  Interventions: Other: olfactory stimulation; Other: functional MRI
- OT non exposed patients (Active Comparator): children non- OT exposed have olfactory test and fMRI
  Interventions: Other: olfactory stimulation; Other: functional MRI

INTERVENTIONS:
Other: olfactory stimulation — the patients have a sniff-test
Other: functional MRI — patients have a an f MRI

SUMMARY:
Studying the cerebral activity of children with Prader-Willi Syndrom (PWS) when the study propose to them nasal activations.

DETAILED DESCRIPTION:
The present study propose to implement fMRI and olfactory tests to describe olfactory brain activation and olfactory skills in early OT-exposed and non-exposed children with PWS.

This study is part of a wider project in collaboration with the team of S. Steculorum at the Max Planck Institute in Germany who assess the architectural and molecular characterization of the olfactory system development in a mice model of PWS and the role of early OT treatment.

Moreover, the study will take advantage of the MRI to document the long-term brain connectivity of early OT-exposed and non-exposed children.

ELIGIBILITY:
Inclusion Criteria:

* child with a genetically confirmed diagnosis of PWS and for whom the genetic subtype (deletion or non deletion) has been identified
* Child aged between 5 and 7 years
* Child with a planned hospitalization at the Toulouse reference center for PWS

Exclusion Criteria:

* Presence of a contraindication to MRI
* Allergy to any of the fragrances used in the olfactory test
* Presence of an ENT infection such as rhinitis or sinusitis on the day of inclusion
* Reported anosmia
* Administrative problems.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
hyperactivation of the right amygdala in young children with PWS not early OT-exposed and aged between 5 and 7 years in response to a sweet food odor compared to a neutral non-food odor. | day 1
  intensity of right amygdala in fMRI

SECONDARY OUTCOMES:
hyperactivation of the right amygdala in PWS children stimulated by a sweet food odor vs. a non-food odor compared to non-exposed children. | day 1
  intensity of right amygdala in fMRI
composite outcome witn an association between olfactory fMRI results and eating behavior in early OT-exposed and non-exposed children with PWS. | day 1
  scores of the eating beahaviour questionnaires
olfactory skills in early OT-exposed and non-exposed children with PWS. | Day 1
  scores of the sniff test between OT-exposed and non-exposed children.
resting brain connectivity in early OT-exposed and non-exposed children with PWS. | day 1
  brain connectivity in fMRI between OT-exposed and non-exposed children.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle DIENE, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No